CLINICAL TRIAL: NCT00212576
Title: Promoting Early School Readiness in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12582; 2R01HD047740-05 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Language Development Disorders
Keywords: Child development; Language Development; Parenting
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Building Blocks (0-3) (Experimental): Randomized at birth to receive Building Blocks Project from birth through 3 years of age.
  Note: This arm not followed past 3 years of age; NOT re-randomized to any group at age 3.
  Interventions: Behavioral: Building Blocks Project
- VIP (0-3), VIP (3-5) (Experimental): Randomized at birth to receive Video Interaction Project from birth through 3 years of age.
  Re-randomized at 3 years to receive Video Interaction Project from 3-5 years of age.
  Interventions: Behavioral: Video Interaction Project
- VIP (0-3), Control (3-5) (Experimental): Randomized at birth to receive Video Interaction Project from birth through 3 years of age.
  Re-randomized at 3 years to receive care as usual (control) from 3-5 years of age.
  Interventions: Behavioral: Video Interaction Project
- Control (0-3), VIP (3-5) (Experimental): Randomized at birth to receive care as usual (control) from birth through 3 years of age.
  Re-randomized at 3 years to receive Video Interaction Project from 3-5 years of age.
  Interventions: Behavioral: Video Interaction Project
- Control (0-3), Control (3-5) (No Intervention): Randomized at birth to receive care as usual (control) from birth through 3 years of age.
  Re-randomized at 3 years to receive receive care as usual (control) from 3-5 years of age.

INTERVENTIONS:
Behavioral: Video Interaction Project — While waiting to see the primary care provider for well child care, the family meets with a child development specialist, who videotapes the parent and infant interacting together. The videotape is then rewound and watched together by the parent and child development specialist. This leads to a discussion about child development, infant cues and parenting, with the child development specialist building on observed strengths in the interaction. In addition, families are provided with parenting pamphlets developed for the project, and with inexpensive developmentally stimulating toys.
  Arms: Control (0-3), VIP (3-5); VIP (0-3), Control (3-5); VIP (0-3), VIP (3-5)
Behavioral: Building Blocks Project — This project employs a public health approach to facilitate parental engagement in child development. Families are sent monthly newsletters that focus on child development, infant cues and parenting; included with each newsletter is an inexpensive, developmentally stimulating toy. In addition, families periodically receive Ages and Stages Questionnaires, which they complete and mail back to the program. Based on the questionnaires, the program determines whether the infant has screened positive for possible developmental delay and provides this information to both the family and the primary care provider.
  Arms: Building Blocks (0-3)

SUMMARY:
This project will measure the degree to which parenting programs based in pediatric primary care can be effective in promoting language development and school readiness in at-risk young children.

The study is a randomized controlled trial in which two different primary care-based parenting programs will be compared to a control group in a population that is at risk on the basis of poverty. The two programs represent varying levels of low intensity, but each has the same goals: enhancing parent-child interaction in order to improve language, cognitive and social-emotional development and ultimately promote school readiness and school performance.

One program is called the "Video Interaction Project". While waiting to see the primary care provider for well child care, the family meets with a child development specialist, who videotapes the parent and infant interacting together. The videotape is then rewound and watched together by the parent (and infant!) and child development specialist. This leads to a discussion about child development, infant cues and parenting, with the child development specialist building on observed strengths in the interaction. In addition, families are provided with parenting pamphlets developed for the project, and with inexpensive developmentally stimulating toys.

The other program is called the "ASQ-Building Blocks Project". This project employs a public health approach to facilitate parental engagement in child development. Families are sent monthly newsletters that focus on child development, infant cues and parenting; included with each newsletter is an inexpensive, developmentally stimulating toy. In addition, families periodically receive Ages and Stages Questionnaires, which they complete and mail back to the program. Based on the questionnaires, the program determines whether the infant has screened positive for possible developmental delay and provides this information to both the family and the primary care provider.

This study will test 2 hypotheses:

1. Primary care based parenting interventions can impact parent-child interaction, early child development and school readiness.
2. Interventions of differing intensity will have impacts of differing magnitude depending on the risk level of the family.

DETAILED DESCRIPTION:
This project will measure the degree to which parenting programs based in pediatric primary care can be effective in promoting language development and school readiness in at-risk young children. The study will represent a collaboration between the Department of Pediatrics at New York University School of Medicine - Bellevue Hospital Center, the Medical and Health Research Association of New York City, Inc., and the Center for Research on Culture, Development and Education at New York University Steinhardt School of Education. Initial funding was provided by NICHD for 4 years. NICHD provided 5 additional years of competing renewal funding beginning in July, 2010.

The study is a randomized controlled trial in which two different primary care-based parenting programs will be compared to a control group in a population that is at risk on the basis of poverty. The two programs represent varying levels of low intensity, but each has the same goals: enhancing parent-child interaction in order to improve language, cognitive and social-emotional development and ultimately promote school readiness and school performance.

One program is called the "Video Interaction Project". While waiting to see the primary care provider for well child care, the family meets with a child development specialist, who videotapes the parent and infant interacting together. The videotape is then rewound and watched together by the parent and child development specialist. This leads to a discussion about child development, infant cues and parenting, with the child development specialist building on observed strengths in the interaction. In addition, families are provided with parenting pamphlets developed for the project, and with inexpensive developmentally stimulating toys.

The other program is called the "ASQ-Building Blocks Project". This project employs a public health approach to facilitate parental engagement in child development. Families are sent monthly newsletters that focus on child development, infant cues and parenting; included with each newsletter is an inexpensive, developmentally stimulating toy. In addition, families periodically receive Ages and Stages Questionnaires, which they complete and mail back to the program. Based on the questionnaires, the program determines whether the infant has screened positive for possible developmental delay and provides this information to both the family and the primary care provider.

The study will take place at Bellevue Hospital Center, a public hospital serving low socioeconomic status families from throughout New York City. Infant-mother dyads will be enrolled during the postpartum period and followed through age 2 years. Periodic assessments will be performed of parent-child interaction and child developmental outcome.

At age 3 years, VIP and control families were re-randomized to receive either additional VIP from age 3 to 5 years or to control during that period. This factorial design will allow for assessment of dose and timing in relation to outcomes.

We further plan to follow children into school, so that we can assess long-term educational outcomes including standardized test scores. Should long-term funding be obtained, we will follow children through high school to assess intervention impacts on graduation rates.

ELIGIBILITY:
Inclusion Criteria:

* Intention to receive primary care in the well-child clinic (FCC or newborn clinic) at Bellevue Hospital Center.
* Intention to remain in the New York City area for at least 3 years.
* Primary caregiver's language is English or Spanish.
* Birthweight 2000gm or higher
* Gestational age 35 weeks or higher

Exclusion Criteria:

* Significant newborn medical complication
* Significant congenital anomaly or syndrome

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Discipline assessed using the Discipline Survey | 6, 14, 24, 36, 54 mos and in 1st grade
  Discipline mediates effects of poverty on social-emotional outcomes (Gershoff, 2007), and attitudes about discipline practices form early in children's lives (Socolar, 1996).
Stress related to interactions and lack of warmth will be assessed using The Parenting Stress Index - Short Form (PSI) | 6, 14, 24, 36, 54 mos and in 1st grade
  Stress related to interactions and lack of warmth mediate effects of poverty on emotional outcomes.
Bayley Scales of Infant and Toddler Development | 14, 24, and 36 mos
  Will assess cognitive development
Woodcock-Johnson III Tests of Cognitive Abilities | 14, 24, and 36 mos
  Will be used to estimate child's cognitive. Four sub-tests will be used: Verbal comprehension (VC) assesses the comprehension knowledge Cattell-Horn-Carroll cognitive factor (Gc); Memory for Words and Auditory Working Memory assess the short term memory CHC factor (Gsm); Visual Matching measures the CHC processing speed factor (Gs).

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Mendelsohn, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Mendelsohn AL, Dreyer BP, Flynn V, Tomopoulos S, Rovira I, Tineo W, Pebenito C, Torres C, Torres H, Nixon AF. Use of videotaped interactions during pediatric well-child care to promote child development: a randomized, controlled trial. J Dev Behav Pediatr. 2005 Feb;26(1):34-41. PMID 15718881
- [Background] Mendelsohn AL, Valdez PT, Flynn V, Foley GM, Berkule SB, Tomopoulos S, Fierman AH, Tineo W, Dreyer BP. Use of videotaped interactions during pediatric well-child care: impact at 33 months on parenting and on child development. J Dev Behav Pediatr. 2007 Jun;28(3):206-12. doi: 10.1097/DBP.0b013e3180324d87. PMID 17565287
- [Background] Berkule SB, Dreyer BP, Huberman HS, Fierman AH, Mendelsohn AL. Attitudes about shared reading among at-risk mothers of newborn babies. Ambul Pediatr. 2007 Jan-Feb;7(1):45-50. doi: 10.1016/j.ambp.2006.10.004. PMID 17261482
- [Background] Mendelsohn AL, Berkule SB, Tomopoulos S, Tamis-LeMonda CS, Huberman HS, Alvir J, Dreyer BP. Infant television and video exposure associated with limited parent-child verbal interactions in low socioeconomic status households. Arch Pediatr Adolesc Med. 2008 May;162(5):411-7. doi: 10.1001/archpedi.162.5.411. PMID 18458186
- [Background] Berkule SB, Dreyer BP, Klass PE, Huberman HS, Yin HS, Mendelsohn AL. Mothers' expectations for shared reading after delivery: implications for reading activities at 6 months. Ambul Pediatr. 2008 May-Jun;8(3):169-74. doi: 10.1016/j.ambp.2008.01.002. Epub 2008 Apr 8. PMID 18501863
- [Background] Green CM, Berkule SB, Dreyer BP, Fierman AH, Huberman HS, Klass PE, Tomopoulos S, Yin HS, Morrow LM, Mendelsohn AL. Maternal literacy and associations between education and the cognitive home environment in low-income families. Arch Pediatr Adolesc Med. 2009 Sep;163(9):832-7. doi: 10.1001/archpediatrics.2009.136. PMID 19736337
- [Derived] Weisleder A, Cates CB, Harding JF, Johnson SB, Canfield CF, Seery AM, Raak CD, Alonso A, Dreyer BP, Mendelsohn AL. Links between Shared Reading and Play, Parent Psychosocial Functioning, and Child Behavior: Evidence from a Randomized Controlled Trial. J Pediatr. 2019 Oct;213:187-195.e1. doi: 10.1016/j.jpeds.2019.06.037. Epub 2019 Aug 6. PMID 31399245
- [Derived] Cates CB, Weisleder A, Berkule Johnson S, Seery AM, Canfield CF, Huberman H, Dreyer BP, Mendelsohn AL. Enhancing Parent Talk, Reading, and Play in Primary Care: Sustained Impacts of the Video Interaction Project. J Pediatr. 2018 Aug;199:49-56.e1. doi: 10.1016/j.jpeds.2018.03.002. Epub 2018 Apr 24. PMID 29703577
- [Derived] Mendelsohn AL, Cates CB, Weisleder A, Berkule Johnson S, Seery AM, Canfield CF, Huberman HS, Dreyer BP. Reading Aloud, Play, and Social-Emotional Development. Pediatrics. 2018 May;141(5):e20173393. doi: 10.1542/peds.2017-3393. Epub 2018 Apr 9. PMID 29632254
- [Derived] Mendelsohn AL, Dreyer BP, Brockmeyer CA, Berkule-Silberman SB, Huberman HS, Tomopoulos S. Randomized controlled trial of primary care pediatric parenting programs: effect on reduced media exposure in infants, mediated through enhanced parent-child interaction. Arch Pediatr Adolesc Med. 2011 Jan;165(1):42-8. doi: 10.1001/archpediatrics.2010.266. PMID 21199979
- [Derived] Mendelsohn AL, Huberman HS, Berkule SB, Brockmeyer CA, Morrow LM, Dreyer BP. Primary care strategies for promoting parent-child interactions and school readiness in at-risk families: the Bellevue Project for Early Language, Literacy, and Education Success. Arch Pediatr Adolesc Med. 2011 Jan;165(1):33-41. doi: 10.1001/archpediatrics.2010.254. PMID 21199978